CLINICAL TRIAL: NCT04492982
Title: Emotion Regulation Interventions for Preventing Collegiate Escalations in Drinking: A Randomized Controlled Trial to Establish Acceptability, Feasibility and Preliminary Efficacy
Brief Title: Emotion Regulation Interventions for Preventing Collegiate Escalations in Drinking
Acronym: PACER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Beth Russell, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R34AA027455-01A1 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-30 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Abuse
Keywords: emotion regulation; alcohol use; college students
MeSH Terms: conditions — Alcoholism; Emotional Regulation; Alcohol Drinking | interventions — Yoga; Self-Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga (Active Comparator): 60 minute sessions of guided yoga in small group format
  Interventions: Behavioral: Yoga
- Distress Tolerance (Active Comparator): 60 minutes sessions of guided didactic distress tolerance skill building in small group format
  Interventions: Behavioral: Distress Tolerance
- Treatment as Usual (No Intervention): Those recruited through Student Health and Wellness will complete the university standard BASICS intervention.

INTERVENTIONS:
Behavioral: Yoga — 1 hour of group format, guided yoga practice
  Arms: Yoga
Behavioral: Distress Tolerance — 1 hour didactic group format, to develop distress tolerance skills
  Other Names: PRISM (Promoting Resilience in Self-Management)
  Arms: Distress Tolerance

SUMMARY:
In the most recent National Survey on Drug Use and Health (NSDUH), college aged respondents between 18 and 25 years old reported the highest alcohol use rates (over 58%) as well as the highest rates of binge drinking of any age group. High alcohol use/abuse in college students is associated with myriad negative consequences, including fatal and nonfatal injuries and overdoses, impaired academic and vocational performance, violence and other crime, legal problems, unintended pregnancies and sexually transmitted diseases, and social problems. The National Comorbidity Survey underscores that use initiated in this period is not just experimental and recreational but may have lasting effects on consumption trajectories: For the majority of adults diagnosed alcohol use disorders, onset occurred during emerging adulthood. During this stage of development, vast changes in emotion regulation (ER) take place, particularly age-related shifts in the strategies used to manage distress that may lead to alcohol use/abuse (i.e., emotion suppression, inhibitory control, and cognitive reappraisal. Substantial evidence suggests that deficits in ER are strongly related to patterns of alcohol use in young adults. In particular, deficits in the self regulation of discomfort and distress, called distress tolerance, predict alcohol use - specifically, motivation and urgency for use, escalations in consumption, and the development of dependence that may be indicative of alcohol use disorders. Emerging adults who turn to alcohol as a way of coping with distressing emotions are most at risk for heavy alcohol use into adulthood and more severe negative alcohol consequences. Given the variable effectiveness of existing approaches for reducing college students' alcohol use, The investigators contend that interventions may be differentially effective depending on individual characteristics. In particular, students with difficulties in managing distress and discomfort may benefit from more intensive interventions that promote effective ER compared to treatment as usual; further, other background characteristics may predict the efficacy and acceptability of each type of ER intervention. In this R34, investigators will test the acceptability/ feasibility and preliminary efficacy of two complementary interventions (Yoga and Distress Tolerance) on preventing alcohol use in a randomized controlled trial of 180 high-risk college students relative to treatment as usual. Investigators will assess participants' alcohol use (self-report and biomarker measures) and emotion regulation (ER) at baseline along with physiological discomfort sensitivity and psychosocial predictors of treatment efficacy over time, including a post-treatment follow-up. Study aims include:

1. Test feasibility/acceptability of two ER interventions among high-risk emerging adults by documenting rates of recruitment, retention, adherence, and satisfaction.
2. Examine trends in intervention acceptability based on baseline characteristics (i.e., associations between participant retention and participant-rated acceptability and age, gender, family characteristics/dynamics, and predispositions to discomfort tolerance).
3. Test preliminary efficacy of the ER interventions on measures of ER and alcohol use. Hypothesis: Participants in both intervention groups will see greater improvements in ER and alcohol use outcomes compared to the TAU control group.

ELIGIBILITY:
Inclusion Criteria:

* Students who report levels of ER difficulties exceeding the mean reported scores on the Difficulties with Emotion Regulation Scale for college students
* Students who screen positive on first 3 items of the AUDIT (called the "AUDIT-C" on which a score of 4 or more for men or 3 or more for women is indicative of hazardous drinking)
* Students with a status as an enrolled student at UCONN with at least a year of on-campus engagement expected before graduation or a commitment to completing all study activities.

Exclusion Criteria:

* Students who are actively psychotic
* Students who have less than a year of on campus engagement expected before graduation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily Drinking Questionnaire | Measured over a 3 month frame, can be used to calculate weekly or daily consumption
  Measures frequency and quantity of alcohol consumption (scores range from 0 to unlimited) where lower scores indicate better outcomes

SECONDARY OUTCOMES:
Distress tolerance scale | Measure authors Simons and Gaher do not specify; PACER will use 90 days
  Measures individual's ability to maintain goal-directed behavior while distressed (scores range from 16 to 80) where higher scores indicate better outcomes
PACER Feasibility - participation | Participation is dichotomously recorded at each engagement opportunity through study completion (up to 8 months)
  Participant participation rates (scores range from 0% to 100%) where higher scores indicate better outcomes
Rates of excessive drinking | 30 days
  Recent reports of heavy (5+ drinks ) in one sitting (scores range from 0 to unlimited) where lower scores indicate better outcomes
CORE survey of substance use | 30 days
  Core frequency measures of substance use from the list of substances, including alcohol, where lower scores indicate better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Beth Russell, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park CL, Russell BS, Fendrich M, Finkelstein-Fox L, Hutchison M, Becker J. Americans' COVID-19 Stress, Coping, and Adherence to CDC Guidelines. J Gen Intern Med. 2020 Aug;35(8):2296-2303. doi: 10.1007/s11606-020-05898-9. Epub 2020 May 29. PMID 32472486